

## University of California, San Diego Consent to Act as a Research Subject

Mechanisms of Affective Touch in Chronic Pain

### Introduction

The rest of the form and asking for your consent to This section provides a summary of important information. and associates are conducting this research provides additional details. Case participate. Laura Dr.

- You can discuss your decision with others (such as family, friends, or another physician). Research is voluntary - whether or not you join is your decision.
  - You can say yes but change your mind later.
- If you say no, we will not hold your decision against you.
- other benefits you may be entitled Your decision will not affect your health care or any to.
- You can say no even if the person inviting you is part of your healthcare team.
  - Please ask questions or mention concerns before, during or after the research.

We will also examine what risk This research will improve our understanding of how touch can interact with pain suffer from chronic pain. Participation in the The purpose of this study is to compare how different types of touch do or do not effect pain n individuals with and without Il not benefit you directly, but may result in new knowledge that may help others perception, and whether this differs in people with chronic pain. factors might explain differences in touch perception between in and health, and whether this differs in people who chronic pain. study wil

During vicodin, oxycontin, hydrocodone, codeine, heroin) and pregnancy (if applicable). If you test sositive for either, you will be dismissed from the study. These test sessions will involve making atings of a variety of painful or non-painful touch stimuli. Each session will last about 1-2 Ip to 20 participants will also be invited to an additional, optional magnetic resonance sessions, we will first administer a urine test for opiates (drugs like morphine, opium, software) to San Diego campus. complete a series of study questionnaires at home (up to 1 hour) prior to coming into the er of the study team will email you a link to REDCap (online survey laboratory. You will then participate in two study sessions on the UC (MRI) session, with similar touch stimuli. mempe imaging vicodin, positive hours. these

of the study are discomfort from the heat and cold water pain The most commonly expected risks of the study are discomfort from the hthat is administered, and becoming bored or upset with the questionnaires.

The most serious risks of the study may include skin burns, which have not been observed at the injury if you receive an MRI and These risks are t properly screened for metal or medical implants in your body. temperatures and time durations used in the study, or serious were not unlikely since we conduct careful screening and you may stop study procedures at any extremely time.

Please feel free to ask Additional, detailed information about this research is provided below. before signing this consent. questions

## and what is the approximate Why have you been asked to participate, how you were selected, study? participants in the 9 number

been asked to participate in this study because you have a diagnosis of Fibromyalgia, at this site There will be approximately 100 participants or you are a healthy control volunteer. You have

# happen to you in this study and which procedures are standard of care and which xperimental What will are

here are some additional details about what will happen to you if you agree to be in this stud In addition to the information at the beginning of this form,

and practice period will be included. If you are not able to follow instructions or rate your sensations on our scales you may be dismissed from the study and compensated only for Session opiates. A training (if scan while receiving these types of respiratory transducer belt will be affixed around your abdomen in order for us to record your respiration rate. You will then receive several types of touch on your arms or legs, including light brushing, deeper pressure, You will receive the same asked to we can test if you are pregnant types of touch from Session 1 in several different combinations, repeated many times, and In the optional MRI session, you will provide a urine sensations on our scales you may be dismissed from the study and compensated only for 1. In Session 2, you will provide a urine sample to test for pregnancy (if applicable) and or unpleasant they feel. You will be All of these procedures are experimental and not for treatment purposes tapping, heat pain, and pain from submerging your hand in cold water. make ratings about how intense or painful and how pleasant or umpleas around your abdomen. In Session 1, you will provide a sample of your urine so that sample to test for pregnancy (if applicable) and have a MRI are taking any opiate medications. A respiratory transducer belt will be affixed will again be asked to make ratings. applicable) and if you touch.

# approximately 3 blocks of testing. In Session 2, there will be approximately 6 blocks of testing Each Session will last approximately 1-2 hours. In Session 1, there will be How much time will each study procedure take and how long will the study last? Each block of sensory testing will take about 5 minutes. In Session 1, there will be

In addition to the risks What risks are associated with this study?

Participation in this study may involve some added risks or discomforts. described at the beginning of this form,

#### Heat Pain Stimuli 1

This is temporary and will Reddening/darkening of the skin may occur with thermal stimulation. not damage the skin.

Cold Water Bath 7)



ice increased heart rate in response to immersing their hand in the cold water. In extremely rare instances, fainting might occur. It is also possible that discomfort and numbness of the hand may occur during and after submerging the hand into the cold water. This is temporary and will not damage the skin. Participants can remove their hand from the cold water in the event they find it intolerable or do not wish to It is possible (although rare) that participants may experien continue.

# 3) Brushing and Pressure

participant's limb, so all participants will be screened to ensure they do not have any signs of skin compression could theoretically dislodge any active blood clots in the clots present. Repeated

#### 4) MR

Persons "squeezeball" that If you cannot tolerate this, the scan implants, pacemakers, or aneurysm clips may not participate. A checklist of excluded metal objects will be presented to you by the MRI technician or study staff prior to the MRI scan. There is no radiation associated with this type of scan. you can squeeze which will subsequently end the scan. During scanning, the MRI machine produces loud noises, so your ears will be protected by plugs or specialized headphones. Pe or body such as cochlear The MRI scan is not associated with any known risks to your health, but you may be uncomfortable because you will be lying in a small space. If you cannot tolerate this will be stopped immediately. In the MRI scanner, we will provide you with a "squee head electronic objects or certain metal objects in The MRI with any

reliable method of birth control while We encourage you to discuss this issue or vasectorny of the partner (with confirmed negative sperm counts) in a monogamous relationship (same partner). participating in this study. Reliable methods of birth control are: abstinence (not having sex), Reproductive Risks: Due to unknown risks and potential harm to the unborn fetus from MRI, careful use of condoms and contraceptives, intrauterine device (IUD), DepoProvera, tubal ligation, active women of childbearing potential must use a An acceptable, although less reliable, method involves the spermicidal foam or gel and/or a cervical cap or sponge. further with your physicians if you have any questions. sexually oral

Due to unknown risks to the fetus, pregnant women are excluded from participation in this study. Because some methods of birth control are not 100% reliable, a urine pregnancy test is required pregnancy assessment for all females at the beginning of the first and second study session and (if you participate in MRI) at the beginning of the fMRI session. at least 10 days from your last normal menstrual period, if you are a sexually active woman of childbearing potential and not using reliable birth control. We will administer a urine based

## 5) Confidentiality

There is a risk that information collected in our study could become known to individuals not involved in our study. Breaches in confidentiality could impact future insurability or employability. However, in our experience, this has not occurred with this type of research.

Because this is a research study, there may be some unknown risks that are currently unforeseeable. You will be informed of any significant new findings.

age 3 of 6

Protections Program
Protections Program
UC San Diego
Approved
Approved
Do not use after 11/25/2020

Are there risks to the reproductive system or a developing fetus?

Due to unknown risks and potential harm to the unborn fetus from MRI, sexually active women of childbearing potential must use a reliable method of birth control if participating in the MRI Because during the MRI Session, if you are a sexually active woman of childbearing potential and not portion of this study. Pregnant women are excluded from participation in this study. Becau some methods of birth control are not 100% reliable, a urine pregnancy test will be required e birth control. using reliabl

If you pregnancy (e.g., late menstrual After you have been enrolled in this study and during the research, pregnancy testing will be If you have a positive pregnancy test, we will withdraw you from the study. period), please contact the study personnel immediately so that we may provide medical (or your partner) become pregnant or if there is any chance assistance and counseling. performed.

# are What

The alternative to not the alternatives to participating in this study?

I have to participate in this study. This is not a treatment study. participating in this study is to not participate. You do not

### can be reasonably expected? benefits What

the investigator(s) may also learn In addition to the benefits listed at the beginning of this form, the investigator(s) more about touch and pain processing and how these may differ in chronic pain.

## you change your mind about participating? ij What happens

you will be requested to inform If you decide that you no longer wish to continue in this study, the investigators and tell us why you are leaving the study.

You will be told if any important new information is found during the course of this study that affect your wanting to continue. may

# Can you be withdrawn from the study without your consent?

You may be withdrawn from the study for the following reasons: your eligibility information changes, or the study physicians Dr. Mark Wallace or Dr. Krishnan Chakravarthy believes that it is in your best medical interest to leave the study. You may also be withdrawn from the study if you do not follow the instructions given you by the study personnel.

# Will you be compensated for participating in this study?

In compensation for your time and travel, you will receive \$60 for intake/Session 1 and \$60 for Session 2 for a total of \$120. The subset of subjects participating in the MRI session will receive he MRI session. \$120 for tl

# any costs associated with participating in this study? Are there

There will be no cost to you for participating in this study.

What if you are injured as a direct result of being in this study?



you are injured as a direct result of participation in this research, the University of California other form of compensation to you if you are injured. You may call the Human Research ections Program Office at 858-246-HRPP (858-246-4777) for more information about this, The University will not provide about your rights as a research subject or to report research-related problems. any medical care you need to treat those injuries. will provide Protections to inquire any

# What about

are Any other software protected encoded to preserve Data and within the medical center. confidentiality. your name physically and pe from ensure will unique identification number and stored separately information. Digital data will be stored on both phys and will only be accessed by study personnel from verto individual participants in reports of this work a HIPPA-compliant fashion will be processed in a information. confidentiality. \$ identifying æ computers All data reference assigned

research study may be presented at scientific or medical meetings or published in scientific journals. Your identity and/or your personal health information will not be disclosed unless it is The results of this safety of yourself or others. always some risk that even de-identified information might be re-identified. Research records will be kept confidential to the extent allowed by law. authorized by you, required by law, or necessary to protect the journals. IS. There

Participant information may be provided to Federal and other regulatory agencies as required. The Food and Drug Administration (FDA), UCSD Institutional Review Board, and NIH, for example, may inspect research records and learn your identity if this study falls within its jurisdiction.

San will be created for you anyway to ensure that this important information is available to doctors in and If you choose to participate in this study, your medical record at the University of California, Diego will indicate that you are enrolled in a research study. Information about the research any medications or devices you are being given as a participant may also be included in your medical record. This part of the medical record will only be available to people who have authorized access to your medical record. If you are not a patient at UCSD, a medical record case of an emergency. medical record.

Certificate may not disclose or use information, documents, or biospecimens that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other action, suit, or proceeding, or be used as evidence unless you have consented for this use. Information, documents, or biospecimens protected by this Certificate cannot be disclosed to anyone else who Researchers with this is not connected with the research unless there is a federal, state, or local law that requires disclosure (such as to report child abuse, elder abuse, intent to hurt self or others, or communicable diseases), you have consented to the disclosure, including for your medical treatment; or it is used for other scientific research, as allowed by federal regulations protecting This research is covered by a Certificate of Confidentiality from NCCIH. research subjects. The Certificate cannot be used to refuse a request for information from personnel of federal or state government agency sponsoring the project that is needed for auditing or program evaluation



You should also understand meet the requirements of the Food and Drug Administration (FDA). You should also understan that a Certificate of Confidentiality does not prevent you from voluntarily releasing information by NCCIH which is funding the project or for information that must be disclosed in order to your research information released to an insurer, medical care provider, or any other person not connected with the research, you must provide consent to allow the research to release it. about yourself or your involvement in this research. If you want

l to in this informed consent document, such as research data entered into your of Confidentiality will not be used to prevent disclosure for any purpose you The Certificate have consented medical record

This Web site will not include information that can identify you. At most, the Web A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required You can search this Web site at any time. site will include a summary of the results. "aw. by U.S.

health information is uncovered such as an unexpected finding on your brain scan, you will be However, if important Will you receive any results from participating in this study?
You will not receive any individual research results from this study. notified.

# Who can you call if you have questions?

If you have other 4968. Case at 858-246 you and your questions have been answered. questions or research-related problems, you may reach Dr. Laura explained to study has been

inquire about your rights as a research subject or to report research-related problems the Human Research Protections Program Office at 858-246-HRPP (858-246 You may call 4777) to

### Signature and Consent Your

copy of this consent document and a copy of the "Experimental Subject's Bill of Rights" to keep. received a You have

Please print a copy of this page at least 18 years old, have read this consent form, and agree to participate in this research study. "You agree" below you are indicating that you are for your records. By clicking

| the person conducting | consent discussion (hard copy only) |
|----------------------------|-------------------------------------|
| Signature of the person of | the informed consent dis |

Date

09/18/2020 11/25/2020 UC San Diego Approved
Current Approval:
Do not use after